CLINICAL TRIAL: NCT05878886
Title: Effect of Mangrove-sword Bean-food Bar on the Weight and Weight-for-Age Z Score of Under-five Children Affected by Landslide Disaster. The Pre-post Intervention Study Towards 34 Under-five Children During 15 Days
Brief Title: Mangrove-sword Bean-food Bar on the Weight and Weight for Age Z Score of Under-five Children
Acronym: MFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fatmah Fatmah, Principal Investigator, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Universitas Indonesia (UI); PUTI Q1 Grants 2023 (Other Grant/Funding Number: University of Indonesia)
Record Dates: First submitted 2023-05-13; First posted 2023-05-26 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Nutrition Poor
Keywords: Older people; under-five children; disaster; weight; mangrove-sword bean-food bar
MeSH Terms: conditions — Malnutrition; Body Weight

STUDY DESIGN:
Intervention Model Description: Treatment group consumed 50 g mangrove sword bean food bar each day during 15 days.
  Control group consumed 50 g sword bean food bar each day during 15 days. Mothers of two groups received balanced nutrition education once at the first week of study.
  The compliance of subject consumed food bar undertaken by home visit of field enumerators to subjects' house.
  They collected three days food recalls and monitored the distribution and stocks of food bar at the subjects' house.
Who Masked: Participant
Masking Description: All subjects at treatment group given mangrove sword bean food bar during 15 days to examine their weight and WAZ score at pre-post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment group received 50 g mangrove sword bean food bar during 15 days.
  Interventions: Dietary Supplement: Emergency Food Product
- Control group (Placebo Comparator): Control group received 50 g sword bean food bar during 15 days.
  Interventions: Dietary Supplement: Emergency Food Product

INTERVENTIONS:
Dietary Supplement: Emergency Food Product — Each subjects of treatment group consumed 50 g food bar during 15 days. Monitoring of compliance undertaken by home visit to recall daily food consumption three days a week and to record the food bar stocks at home during study, and also weekly weight measurement.
  Other Names: Mangrove sword bean food bar

SUMMARY:
The goal of this clinical trial is to assess the effect of the food bar made from api-api mangrove (Avicennia marina) and sword bean (Canavalia ensiformis) blends on the weight and Weight-for-Age Z score affected by a landslide disaster.

The main questions aimed to answer are:

* Food bar supplementation can effect the weight and WAZ score of under-five children affected by landslides disaster?
* Balanced nutrition education can increase the mothers' knowledge on the balanced nutrition of under-five children?

Participants divided in to two group i.e.:

* Treatment/intervention group consumed 50 g mangrove sword bean food bar each day during 15 days.
* Control group consumed 50 g sword bean food bar each day during 15 days.
* Each group received balanced nutrition for mothers once at the first week of study.

DETAILED DESCRIPTION:
Eligibility Criteria for Under-five children:

* Aged between 12 and 59 months
* Male and female
* Living in Cihanjuang Village of Sumedang District which affected by the landslide disaster
* Had malnutrition, normal, or over-nutrition status, and not suffering from infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 59 months
* Male and female living in Cihanjuang Village of Sumedang District who affected by the landslide disaster
* Had malnutrition, normal, or over-nutrition status
* Not suffering from infectious diseases
* Willing to avoid consumption of any snacks other than the food bars and plain water

Exclusion Criteria:

* Suffered from infectious or chronical diseases

Ages: 12 Months to 49 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Effect of mangrove-sword bean-food bar on the weight and Weight-for-Age Z score (WAZ) of under-five children affected by landslide disaster | Two weeks
  Change of weight measured by digital weighing. Change of Weight for Age Z score measured by using Nutri Survey Software. Mean difference of weight and Weight-for-Age Z score were calculated as the value at two weeks minus the value at baseline.

SECONDARY OUTCOMES:
Change of mothers' balanced nutrition knowledge | Two weeks
  Knowledge score of mothers of underfive children on the balanced nutrition at pre-post study measured by baseline and end-line questionnaires.
  Mean difference of balanced nutrition knowledge of mothers was calculated as the value at two weeks minus the value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Fatmah Fatmah, Dr, Principal Investigator — UI
Locations (1):
- Cihanjuang Village, Sumedang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No